CLINICAL TRIAL: NCT03673033
Title: Can the Effects of Cold and Hot Ischemia Time on Biliary Complications in Live Donor Liver Transplantation Be Classified?
Brief Title: Biliary Complications in Live Donor Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, cihan gokler, Principal invastigator, Inonu University
Other Study IDs: 2018/18
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2018-09

CONDITIONS: Biliary Stricture; Bile Duct Stenosi; Bile Leak; Bile Duct Injury
Keywords: Transplantation, Hepatic, Cirrhosis, Bile duct
MeSH Terms: conditions — Fibrosis | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: liver transplantation — calculation of hot and cold ischemia durations from donor artery cut-off time in liver transplantation

SUMMARY:
The study was designed as a prospective cohort study. The effects of hot and cold ischemic times during live donor liver transplantation on postoperative 1-3 and 6 month follow up biliary complications will be investigated.

DETAILED DESCRIPTION:
The invastigators will record the age, gender, weight, diagnosis, presence of hcc (hepatocellular carcinoma), whether transcatheter embolization (transarterial radiolabelization) is performed, meld score, age of donor, gender, graft hepatic artery diameter, bile duct diameter and number before surgery.

During the operation,

The duration of ischemia will be evaluated as three stages.

During the first stage donor hepatectomy, the time from the interruption of the hepatic artery to the first administration of the solution to the bile ducts on the back table will be recorded and recorded as the first ischemia time.

The time from the administration of the solution to the biliary system on the stage 2 back-to-back table until the cold anastomosis is performed will be recorded as the duration of cold ischemia.

The time from the third graft to receipt of the graft to the end of the hepatic artery anastomosis will be recorded as the second ischemia time.

The duration of operation, whether or not pringle maneuvers were performed, hepatic artery thrombus, graft bile number, number of bile anastomoses, lowest biliary tract diameter and hepatic artery diameter

After the surgery,

The use of immunosuppression (Tacrolimus, certican or combined use) will be recorded.

During the follow-up period of 1,3,6 months, complaints of the patients, laboratory values and imaging methods as well as whether or not there is biliary complication (leakage, stenosis) will be recorded.

If the complication develops during follow-up, the procedure (follow-up, ercp, ptk, surgery) will be recorded.

Since the study is observational, normal treatment will not be involved.

Participants will not be included in the study in the presence of hepaticojejunostomy patients, cadaveric transplant patients, pediatric transplant patients, Cmv infection, hepatic artery thrombosis, portal thrombosis, acute rejection in the first operation.

Participants with live donor liver transplant patients, multiple gallbladder anastomoses or single bile duct multiple anastomoses will be included.

When the power analysis for the study was taken as α = 0.05 and 1-β (power) = 0,80, it was calculated that at least 99 patients should be taken to have a difference of 38% in the rates of biliary complication in cold ischemia.

The demographic and all findings of the disease will be collected at excell and at the end of the study all the findings will be statistically evaluated and the results will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Live donor liver transplantation Emergency Live donor liver transplantation Multiple or single bile duct anastomosis in liver transplantation

Exclusion Criteria:

Hepaticojejunostomy Cadaveric liver transplantation Pediatric liver transplantation Cmv infection presence Hepatic arterial thrombus Porta thrombus Acute rejection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with live donor liver transplant for any reason
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-03 (Actual)

PRIMARY OUTCOMES:
development of biliary complication in the first month after liver transplantation | 1 month
  biliary complication at the first month after transplantation and whether this complication is interfered with or not will be evaluated.

SECONDARY OUTCOMES:
development of biliary complication in the three months after liver transplantation | 3 months
  biliary complication at the third month after transplantation and whether this complication is interfered with or not will be evaluated.
development of biliary complication in the six month after liver transplantation | 6 months
  biliary complication at the sixth month after transplantation and whether this complication is interfered with or not will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Cihan Gokler, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
de-identified individual participant data for all primary, secondary and tertiary outcome measures will be made available
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: data will be available within 6 months of study completion
Access Criteria: data access request will be reviewed by an external independent review panel.